CLINICAL TRIAL: NCT05721196
Title: Culturally Adapted Psychoeducation (CaPE) for Bipolar Disorders in Nigeria: A Pilot Randomised Controlled Trial
Brief Title: Culturally Adapted Psychoeducation (CaPE) for Bipolar Disorders in Nigeria
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nottingham Trent University (Other)
Collaborators: University of Toronto (Other); Teesside University (Other); University of Manchester (Other)
Responsible Party: Principal Investigator, Dr Dung Jidong, PhD, Principal Investigator, Nottingham Trent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0000-0001-5034-0335e
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culturally adapted Psychoeducation (CaPE) (Experimental)
  Interventions: Behavioral: Culturally adapted Psychoeducation (CaPE)
- Treatment as Usual (TaU) (Active Comparator)
  Interventions: Drug: Treatment as Usual (TaU)

INTERVENTIONS:
Behavioral: Culturally adapted Psychoeducation (CaPE) — This intervention consisted of 12 psychoeducation sessions, one session per week, that would be administered on an individual patient basis and to be added to treatment as usual. Each session lasted for approximately 1 h, beginning with a 20-30 min presentation on the topic of the day, followed by a related exercise (e.g., drawing a life chart or compiling a list of potential triggers for relapse). The content is a reduced and modified version of the Barcelona Psychoeducation Program for bipolar disorders.
  Arms: Culturally adapted Psychoeducation (CaPE)
Drug: Treatment as Usual (TaU) — This group of patients will receive routine treatment, which in Nigeria means attending the outpatient clinic and taking prescribed medication.
  Arms: Treatment as Usual (TaU)

SUMMARY:
Bipolar disorders are chronic mental health disorders that often result in functional impairment, constituting a significant disease burden. It also accounts for seven per cent of disability-adjusted life years caused by mental disorders. Four out of ten persons with a probable diagnosis of bipolar disorders received no mental health care within the preceding twelve months. Compared to the general population, individuals with bipolar disorders tend to have a significantly higher rate of associated suicide mortality. Within the last decade, these mortality rates have substantially increased, suggesting the need for targeted research to address the unresolved needs of individuals suffering from bipolar disorders. A recent meta-analysis found that compared to the general population, bipolar patients had reduced life expectancy with about thirteen years of potential life loss.

Bipolar disorders are historically under-researched compared to other mental health disorders, especially in Sub-Saharan Africa and Nigeria. Our recent study on bipolar disorders in Nigeria provided insight into contextual knowledge and beliefs about bipolar disorders, including the lived experiences of patients with bipolar disorders, their caregivers, and clinicians in Nigeria. The study recommended culturally adapted psychosocial intervention for bipolar patients, hence the proposed research.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of DSM IV bipolar affective disorder
* currently euthymic (BDI < 12 and YMRS < 8)
* age 18-65 years, participants engaged with the mental health services for the preceding 6 months
* able to give written informed consent
* resident of the trial catchment area and
* the ability to speak English.

Exclusion Criteria:

* severe cognitive impairment
* currently experiencing relapse (mania, hypomania, mixed or depressive)
* being actively suicidal
* the presence of any comorbid psychiatric illness such as substance misuse or alcohol dependence according to DSM IV criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Pain reduction | Change is being assessed at baseline, at 12 weeks end of intervention, at 3-months, and at 6-months post-intervention
  Patients' pain reduction would be assessed by the Visual Analogue Scale. For example, 0 = No pain and 10 = worst pain.

SECONDARY OUTCOMES:
Bipolar knowledge and attitude | Change is being assessed at baseline, at 12 weeks end of intervention, at 3-months, and at 6-months post-intervention
  Bipolar knowledge and attitude would be assessed using the Bipolar Knowledge & attitude questionnaire
Medication adherence | Change is being assessed at baseline, at 12 weeks end of intervention, at 3-months, and at 6-months post-intervention
  Medication adherence would be assessed using the Morisky measure of medication adherence survey
Severity of mood symptoms | Change is being assessed at baseline, at 12 weeks end of intervention, at 3-months, and at 6-months post-intervention
  Severity of mood symptoms would be assessed using the Young Mania Rating Scale (YMRS) or Beck's Depression Inventory
Quality of life | Change is being assessed at baseline, at 12 weeks end of intervention, at 3-months, and at 6-months post-intervention
  Quality of life would be assessed using the Health-related quality of life was also measured using EuroQoL (EQ-5D)

IPD SHARING:
Plan to Share IPD: Yes